CLINICAL TRIAL: NCT06461650
Title: Preoperative Nicotine Cessation for Women With Breast Cancer Recommended for Reconstruction
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UF-BRE-013; IRB202401102 (Other: University of Florida)
Record Dates: First submitted 2024-06-11; First posted 2024-06-17 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Breast Cancer
Keywords: breast cancer; nicotine cessation; mastectomy; reconstruction; smokers
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nicotine cessation program (Experimental)
  Interventions: Behavioral: Nicotine cessation program

INTERVENTIONS:
Behavioral: Nicotine cessation program — Participants will complete up to 4 sessions of a nicotine cessation program over either 12-24 weeks if receiving neoadjuvant therapy (i.e. chemotherapy or hormonal/endocrine therapy) prior to surgery or over 4-6 weeks if not receiving neoadjuvant therapy prior to surgery. Each session will be 30-60 minutes long. Participants receiving neoadjuvant therapy will also be eligible for nicotine replacement therapy; however, it must be stopped 6 weeks before surgery.

SUMMARY:
Close to 20% of cancer patients currently use nicotine products. Nicotine use in breast cancer patients is associated with poorer overall outcomes, including worsened survival and increased surgical complications. Nicotine cessation is rarely addressed in breast cancer patients at the time of diagnosis and may be a missed opportunity to optimize patient outcomes. Patients that use nicotine products are not offered reconstruction at time of mastectomy or oncoplastics at the time of lumpectomy, which can be emotionally distressing in women with breast cancer. Reconstruction could be an additional motivating factor in nicotine cessation success.

This study aims to evaluate the feasibility of a nicotine cessation program designed by Area Health Education Center (AHEC) in the target population. The study is designed to test the acceptability, and preliminary efficacy of a formal nicotine cessation program in women actively using nicotine products with breast cancer recommended for reconstructive or oncoplastics surgery.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥ 18 years of age and ≤ 80 years of age.
* Women who are diagnosed with Stage 0 - 3 breast cancer confirmed by biopsy
* Women who have been recommended to have reconstruction at time of mastectomy or oncoplastics at time of lumpectomy
* Participants who actively use nicotine products defined as any self-reported nicotine use within the past month
* Participant agrees to comply with all the study-related procedures.

Exclusion Criteria:

* Patients not eligible for reconstruction or oncoplastics for other reasons including BMI>35 or inflammatory breast cancer or based on surgeon discretion.
* Prisoners or subjects who are involuntarily incarcerated, or subjects who are compulsorily detained for treatment of either a psychiatric or physical illness.
* Patients unable to complete the sessions because of language, travel or technology barriers
* Patients already actively participating in another cessation program
* Patients who are pregnant.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-11-14 (Actual); Primary Completion 2028-03 (Estimated); Study Completion 2029-03 (Estimated)

PRIMARY OUTCOMES:
Feasibility | 12-24 weeks (if receiving neoadjuvant therapy prior to surgery) or 4-6 weeks (if not receiving neoadjuvant therapy prior to surgery)
  Determine the feasibility of the nicotine cessation program used in this study, as measured by subject participation in at least one program session after study enrollment.

SECONDARY OUTCOMES:
Acceptability | 10-30 weeks
  Determine the acceptability of the nicotine cessation program used in this study, as measured by participant surveys administered at baseline, at completion of the nicotine cessation program sessions, and at 6 weeks postoperatively.
Preliminary efficacy | 10-30 weeks
  Determine the preliminary efficacy of the nicotine cessation program used in this study, as measured by participant surveys administered at baseline, at completion of the nicotine cessation program sessions, and at 6 weeks postoperatively.
Short-term impact on nicotine cessation | 10 days prior to surgery
  Determine the short-term impact on nicotine cessation of the nicotine cessation program used in this study, as measured by cotinine levels prior to surgery.
Long-term impact on nicotine cessation | 12 months postoperatively
  Determine the long-term impact on nicotine cessation of the nicotine cessation program used in this study, as measured by a participant survey administered 12 months postoperatively.
Patient engagement | 12-24 weeks (if receiving neoadjuvant therapy prior to surgery) or 4-6 weeks (if not receiving neoadjuvant therapy prior to surgery)
  Determine patient engagement, as measured by number of program sessions completed and which program sessions were completed.
Surgical procedure | At surgery
  Determine the surgical procedure each participant underwent following completion of the nicotine cessation program, including if the participant had either reconstruction or oncoplastics at the time of this surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Fieber, MD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States